CLINICAL TRIAL: NCT04336293
Title: sTMS for Substance Use-disordered Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: D3338-P; RX003338 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2020-03-20; First posted 2020-04-07 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cocaine Addiction; Opioid Addiction; Alcohol Addiction
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: double blind, sham controlled RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active (Experimental): active sTMS
  Interventions: Device: sTMS
- sham (Sham Comparator): sham sTMS
  Interventions: Device: sham sTMS

INTERVENTIONS:
Device: sTMS — sTMS will be delivered following NeoSync guidelines using the device user
  manual
  Arms: active
Device: sham sTMS — sham sTMS will be delivered following NeoSync guidelines using the device user manual
  Arms: sham

SUMMARY:
The purpose of this study is to determine if synchronized transcranial magnetic stimulation is safe and tolerable in individuals with cocaine, opioid, or alcohol use disorders.

DETAILED DESCRIPTION:
All non-life-saving human research studies suspended by sponsor in response to COVID19 social distancing policies

The goal of this proposal is to evaluate preliminary participant response to a pilot, controlled, feasibility study to evaluate changes in craving, substance use, and quality of life after 6 weeks of a low-risk non-invasive brain stimulation technique, called Synchronized Transcranial Magnetic Stimulation (sTMS), compared to sham, in Veterans with a substance use disorder (SUD). An important focus of this application will be evaluating the acceptability, tolerability, and safety of sTMS in this population. To the investigators knowledge, sTMS has never been used for SUDs, and holds considerable promise as a future treatment option for these prevalent disorders. However initial work in the acceptability, tolerability, and safety of this approach must be conducted first. This project is the first step towards the investigators long-term goal, which is to combine non-invasive brain stimulation with individualized psychotherapy or pharmacotherapy to reduce SUD problems and improve quality of life for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Eligible male and female Veterans
* between ages 18-70,
* Veterans who currently meet criteria for SUD, and, if applicable, have stable treatment regimen (i.e., medications and/or therapy) for at least 6 weeks prior to study procedures
* ongoing medications and psychotherapy will be allowed to continue unchanged during the study
* for safety, participants must also meet established criteria for MRI exposure, which is implemented as a conservative measure given the novel application of sTMS in this population

Exclusion Criteria:

* pregnancy/lactation,
* history of moderate or severe traumatic brain injury,
* current or prior neurologic disorder or lifetime history of

  * seizure disorder
  * CNS tumors
  * stroke
  * cerebral aneurysm,
* unstable medical condition,

  * active suicidality as assessed with the Columbia-Suicide Severity Rating Scale
  * primary psychotic disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) | 6 weeks
  Quality of Life Enjoyment and Satisfaction Questionnaire
  The Q-LES-Q-SF evaluates general activities that are assessed in the longer form of the Q- LES-Q. Each item uses a 5-point scale ranging from 1 (very poor) to 5 (very good). A total score is derived from 14 items with a maximum score of 70 and with higher scores indicating greater life satisfaction and enjoyment.
substance specific craving | 6 weeks
  self reported reactivity to associated cues with 8 items ranked 1-7--higher scores indicating greater craving/urges
Social and Occupational Functioning Assessment Scale (SOFAS) | 6 weeks
  The SOFAS is a global rating of current functioning ranging from 0 to 100, with lower scores representing lower functioning.

CONTACTS AND LOCATIONS:
Overall Officials: John E McGeary, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jampel J, Quinn MJ, Catalano JL, Benca-Bachman CB, Brick L, Philip NS, Swift RM, McGeary JE. Synchronised transcranial magnetic stimulation for substance use-disordered Veterans: protocol for the pilot sham-controlled acceptability trial. BMJ Open. 2023 Jan 30;13(1):e066175. doi: 10.1136/bmjopen-2022-066175. PMID 36717148

DOCUMENTS (1):
  • Informed Consent Form (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04336293/ICF_000.pdf